CLINICAL TRIAL: NCT03400722
Title: Double Ovarian Stimulation as Accumulation Strategy for Older Infertile Patients With Suboptimal Ovarian Response in Assisted Reproductive Treatment
Brief Title: Double Ovarian Stimulation as Accumulation Strategy for Older Infertile Patients With Suboptimal Ovarian Response
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Nova Clinic, Russia (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: NCT 03230763
Record Dates: First submitted 2017-12-19; First posted 2018-01-17 (Actual); Last update posted 2018-01-17 (Actual); Status verified 2018-01

CONDITIONS: Infertility, Female; Ovarian Stimulation; In Vitro Fertilisation
Keywords: Suboptimal ovarian response; Ovarian Stimulation; Infertility, Female; In Vitro Fertilisation
MeSH Terms: conditions — Infertility, Female | interventions — pergoveris; Clomiphene

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- DUOSTIM group (Experimental): Pergoveris 150 -300 IU start from day 2 of the cycle up to the day of trigger, GnRH antagonist 0,25 mg start from day 7-8 of the cycle up to the day of trigger, final trigger of ovarian stimulation - GnRH-a 0,2 mg, oocyte retrieval 35 hours after trigger, stop period for 5 days, after stop period start Pergoveris 150 - 300 IU start up to the day of trigger, GnRH antagonist 0,25 mg start from day 6 of ovarian stimulation up to the day of trigger, final trigger of ovarian stimulation - GnRH-a 0,2 mg, oocyte retrieval 35 hours after trigger. After oocyte retrieval fertilization will be carried out by IVI or ICSI, the development of embryos will be carried out up to blastocyst stage, then blastocyst vitrification will be performed.
  Interventions: Drug: Pergoveris
- Modified Shanghai Protocol group (Experimental): Clomiphene 50 mg start from day 2-3 of the cycle up to the day of trigger, Pergoveris 150 - 300 IU - 6,8, 10 days of the cycle, final trigger of ovarian stimulation - GnRH-a 0,2 mg, oocyte retrieval 35 hours after trigger, after stop period for 2-3 days start Pergoveris 150 - 300 IU up to the day of trigger, final trigger of ovarian stimulation - GnRH-a 0,2 mg, oocyte retrieval 35 hours after trigger. After oocyte retrieval fertilization will be carried out by IVI or ICSI, the development of embryos will be carried out up to blastocyst stage, then blastocyst vitrification will be performed.
  Interventions: Drug: Clomiphene

INTERVENTIONS:
Drug: Pergoveris — Two controlled ovarian stimulation within the same menstrual cycle. It will be followed by ovarian puncture, fertilisation of oocyte by IVI or ICSI, blastocyst vitrification. If there are 3-5 blastocysts, the embryo accumulation process will be completed and the unfrozen embryos transferred.
  Other Names: antagonist of gonadotropin releasing hormone; agonist of gonadotropin releasing hormone
  Arms: DUOSTIM group
Drug: Clomiphene — Two controlled ovarian stimulation within the same menstrual cycle. It will be followed by ovarian puncture, fertilisation of oocyte by IVI or ICSI, blastocyst vitrification. If there are 3-5 blastocysts, the embryo accumulation process will be completed and the unfrozen embryos transferred.
  Other Names: Pergoveris; agonist of gonadotropin releasing hormone
  Arms: Modified Shanghai Protocol group

SUMMARY:
Patients with infertility of the older age group of 37-42 years - a large cohort of patients of reproductive medicine. Two possible causes reduce their probability of pregnancy - an increasing age and a decrease of the ovarian reserve. In these conditions, the early receipt of embryos for future transfer can serve as a correct strategy for treating infertility in this category of patients. According to statistical data, patients of the 37-42-year-old age group need 3-5 blastocysts, out of them 1-2 euploid to achieve pregnancy.

The POSEIDON group of researchers identified a group of 2b patients with a suboptimal response to the induction of superovulation in IVF programs - patients older than 35 years with a normal ovarian reserve (the number of antral follicles greater than 5 and Anti-Müllerian hormone (AMH) greater than 1.2 ng / ml), resulting in 4-9 oocytes after a standard ovarian stimulation.

In this situation standard stimulation protocols can stretch the process of obtaining embryos indefinitely, during which the patient will move to another age category with a decrease in the likelihood of pregnancy.

Thus, these patients are shown the fastest reception of oocytes and the accumulation of embryos, which can be done using double ovarian stimulation in the same menstrual cycle.

The aim of the study is to compare the different schemes of double stimulation in patients with infertility of the older age group of 37-42 years with the preceding suboptimal response.

Group 1 - patients of the DUOSTIM group. Group 2 - Patients of the Shanghai Protocol.

The investigated parameters - primary outcome measures: total number of retrieved oocytes per cycle, secondary outcome measures: total number of blastocyst per cycle, number of cycles with double ovarian stimulation required to obtain 3-5 blastocyst, time until embryo transfer, pregnancy rate and birth rate This is a prospective randomized non-blinded clinical study.

DETAILED DESCRIPTION:
The aim of the study is to compare the different schemes of double stimulation in patients with infertility of the older age group of 37-42 years with the preceding suboptimal response.

Materials and methods. Patients with preserved ovarian reserve of 37-42 years old, who had the history of standard stimulation in IVF programs, which produce less 4-7 oocytes. Patients will be randomised in two groups. Group 1 - patients of the double ovarian stimulation in the same cycle with recombinant gonadotropin (DUOSTIM group). Group 2 - patients of the double ovarian stimulation in the same cycle with clomifen and recombinant gonadotropin (modified Shanghai Protocol).

The stimulation protocol in the Group 1 - Follitropin and Lutropin Alfa (Pergoveris) 150 -300 IU start from day 2 of the cycle up to the day of trigger, gonadotropin-releasing hormone (GnRH) antagonist 0,25 mg start from day 7-8 of the cycle up to the day of trigger, final trigger of ovarian stimulation - gonadotropin-releasing hormone agonist (GnRH-a) 0,2 mg, oocyte retrieval 35 hours after trigger, stop period for 5 days, after stop period start Pergoveris 150 - 300 IU start up to the day of trigger, GnRH antagonist 0,25 mg start from day 6 of ovarian stimulation up to the day of trigger, final trigger of ovarian stimulation - GnRH-a 0,2 mg, oocyte retrieval 35 hours after trigger.

After oocyte retrieval fertilization will be carried out by invitro insemination (IVI) or intracytoplasmic sperm injection (ICSI), the development of embryos will be carried out up to blastocyst stage, then blastocyst vitrification will be performed. The cycles of double ovarian stimulation will be performed until the patient will have not less than 3-5 blastocysts. Then the embryo accumulation process will be completed and the unfrozen embryos transferred in the hormonal replacement cycle or natural ovulatory cycle.

The stimulation protocol in the Group 2 - Clomiphene 50 mg start from day 2-3 of the cycle up to the day of trigger, Pergoveris 150 IU - 6,8, 10 days of the cycle, final trigger of ovarian stimulation - GnRH-a 0,2 mg, oocyte retrieval 35 hours after trigger, after stop period for 2-3 days start Pergoveris 150 - 300 IU up to the day of trigger, final trigger of ovarian stimulation - GnRH-a 0,2 mg, oocyte retrieval 35 hours after trigger. After oocyte retrieval fertilization will be carried out by IVI or ICSI, the development of embryos will be carried out up to blastocyst stage, then blastocyst vitrification will be performed. The cycles of double ovarian stimulation will be performed until the patient will have not less than 3-5 blastocysts. Then the embryo accumulation process will be completed and the unfrozen embryos transferred in the hormonal replacement cycle or natural ovulatory cycle.

ELIGIBILITY:
Inclusion Criteria:

1. 37 - 42 years of age
2. BMI 18-30 kg\m2
3. Suboptimal ovarian responders with normal ovarian reserve: the number of antral follicles greater than 5 and AMH greater than 1.2 ng / ml, resulting in 4-9 oocytes after a standard ovarian stimulation, according Poseidon classification - group 2b
4. Informed consent

Exclusion Criteria:

1. Medical contraindications for IVF
2. Basal follicle stimulating hormone (FSH) more 15 IU/L
3. Severe mail factor

Ages: 37 Years to 42 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 120 (Estimated)
Dates: Start 2017-12-01 (Actual); Primary Completion 2018-08-01 (Estimated); Study Completion 2019-05-01 (Estimated)

PRIMARY OUTCOMES:
Total number of retrieved oocytes per cycle | up to 9 months
  evaluation the total number of retrieved oocytes after double ovarian stimulation in one cycle

SECONDARY OUTCOMES:
total number of blastocyst per cycle | up to 9 months
  evaluation the total number of blastocyst after double ovarian stimulation in one cycle
Time until embryo transfer | up to 9 months
  period from start double ovarian stimulation until embryo transfer
number of cycles need to treat | up to 9 months
  number of cycles with double ovarian stimulation required to obtain 3-5 blastocyst
pregnancy rate | up to 9 months
  pregnancy rate after embryo transfer of thawed blastocyst
the birth rate | up to 18 months
  the birth rate after embryo transfer

CONTACTS AND LOCATIONS:
Overall Officials: Konstantin Dancheev, Study Director — MEDINSERVIS LLC NOVA CLINIC
Locations (1):
- Irina Zorina, Moscow, Russia

IPD SHARING:
Plan to Share IPD: Undecided